CLINICAL TRIAL: NCT00904618
Title: Better Short-Term Outcomes With The 'U-Method' Compared to the 'Hammock' Technique for the Implantation of the TVT-SECUR Under Local Anesthesia
Brief Title: Safety and Efficacy Study on the Implantation of the Tension-Free Vaginal Tape (TVT-Secur) Under Local Anesthesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: Le-Mai Tu, Centre Hospitalier Universitaire de Sherbrooke
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USherbrooke-001
Record Dates: First submitted 2009-03-11; First posted 2009-05-19 (Estimated); Results first posted 2009-05-19 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2009-04

CONDITIONS: Urinary Stress Incontinence
Keywords: Suburethral slings; Urethra; Urinary incontinence; Urinary stress incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence | interventions — Anesthesia, Local; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TVT-SECUR (Experimental): This study arm consisted of 48 women operated from January 2007 to October 2008. All patients underwent the implantation of the TVT-SECUR for the treatment of stress urinary incontinence or stress predominant mixed urinary incontinence. The surgery was done under local anesthesia by one high-volume surgeon.
  Interventions: Procedure: TVT-SECUR - 'Hammock' technique; Procedure: TVT-SECUR - 'U-Method'; Drug: Local anesthesia (30 to 40 ml of a mixture of 35 ml of lidocaine 2% and 5 ml of bicarbonate 3%).

INTERVENTIONS:
Procedure: TVT-SECUR - 'Hammock' technique — The surgery was done under local anesthesia by one high-volume surgeon. The 'Hammock' technique, similar to the transobturator tape dissection, was used in the first 23 cases and the 'U-Method', similar to the retropubic tape dissection, in the last 25 cases. Interim analysis performed after 23 cases led us to change the technique to the 'U-Method'.
Procedure: TVT-SECUR - 'U-Method' — The surgery was done under local anesthesia by one high-volume surgeon. The 'Hammock' technique, similar to the transobturator tape dissection, was used in the first 23 cases and the 'U-Method', similar to the retropubic tape dissection, in the last 25 cases. Interim analysis performed after 23 cases led us to change the technique to the 'U-Method'.
Drug: Local anesthesia (30 to 40 ml of a mixture of 35 ml of lidocaine 2% and 5 ml of bicarbonate 3%). — Local anesthesia consisted of 30 to 40 ml of a mixture of 35 ml of lidocaine 2% and 5 ml of bicarbonate 3%. Sedation was used in association with local anesthesia, including 1 mg of lorazepam sublingual as well as a combination of 0.5 to 2 mg intravenous (IV) of midazolam and 50 to 200 ug IV of fentanyl. Postoperative analgesia consisted of a prescription of 30 tablets of morphine 5 mg.

SUMMARY:
The objective was to observe the satisfaction of local anesthesia during the implantation of the TVT-SECUR for the treatment of stress urinary incontinence, with the use of questionnaires completed by the patients, and to evaluate the short-term efficacy and safety of the sling, with a comparison of the two techniques of implantation: the 'U-Method' and the 'Hammock' technique.

DETAILED DESCRIPTION:
Stress urinary incontinence (SUI) is a common problem, affecting women of all ages. Treatment options for SUI include physiotherapy and surgical interventions, such as retropubic operations and midurethral slings. Conventional retropubic and transobturator tapes are the preferred choice for most surgeons, because of their wide applicability, technical simplicity and clinical efficacy. The retropubic tape has been effective for many years, but exposes the patients to serious complications, such as bladder perforations, principally because of the use of the retropubic space for the fixation of the tape. In an attempt to avoid the retropubic space, the second generation of slings, the transobturator tape, was introduced. However, prolonged postoperative groin pain as well as vascular injuries have been reported.

The last generation of midurethral slings, the tension-free vaginal tape system (TVT-SecurTM, Gynecare, Ethicon, Somerville, NJ, USA), introduced in 2005, attempts to lower the number of complications, by involving only a small vaginal incision and no exit wound. This 8-cm long laser-cut polypropylene mesh can potentially be implanted under local anesthesia, because of a less-invasive technique using minimal vaginal dissection as well as avoidance of retropubic space and obturator fossa. In the case of conventional midurethral slings, even if their implantation under local anesthesia has been studied and proven relatively safe, this practice has not gained popularity.

This was a prospective, clinical study with primary objective to observe the satisfaction of local anesthesia during the implantation of the TVT-SECUR, with the use of questionnaires completed by the patients. The secondary objective was to observe the short-term efficacy and safety of the sling. The final objective was to compare the two techniques of implantation: the 'U-Method' and the 'Hammock' technique.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stress urinary incontinence or stress predominant mixed urinary incontinence
* Acceptance of local anesthesia

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Le-Mai Tu, MD, MSc, FRCS, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: January 2007 to October 2008 at Centre Hospitalier Universitaire de Sherbrooke (CHUS)
Period: Overall Study
Arm/Group | TVT-SECUR
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TVT-SECUR
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 58 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 0
Region of Enrollment [Number; unit: participants]
  Canada | 48

OUTCOME MEASURES:

1. Primary Outcome: Local Anesthesia Satisfaction
Description: Local anesthesia satisfaction was assessed with a questionnaire completed by the patients. The patients were asked if they would recommend this type of anesthesia (yes or no).
Time Frame: Questionnaire filled 1 week after surgery
Population: 2 patients did not fill out the questionnaire 1 week after surgery
Measure: Number; unit: participants
Arm/Group | TVT-SECUR
Number analyzed (Participants) | 46
participants
  Yes | 43
  No | 3

2. Secondary Outcome: Improvement in Stress Urinary Symptoms.
Description: A questionnaire with a Likert scale from one to five was used to assess the improvement in stress urinary symptoms at six months for each technique, the 'Hammock' technique and the 'U-Method' (1-Worst, 2-Same, 3-Improved, 4-Almost cured, 5-Cured). Patients had to answer 3 or more on the scale to be considered improved.
Time Frame: Six months
Population: The 'Hammock' technique, similar to the transobturator tape dissection, was used in the first 23 cases and the 'U-Method', similar to the retropubic tape dissection, in the last 25 cases. Seven patients for the 'Hammock' technique and three patients for the 'U-Method' did not fill out the questionnaire at six months.
Measure: Number; unit: participants
Groups:
- 'Hammock' Technique: The 'Hammock' technique is similar to the transobturator tape dissection.
- U-Method: The U-Method is similar to the retropubic tape dissection
Arm/Group | 'Hammock' Technique | U-Method
Number analyzed (Participants) | 16 | 22
participants
  Improved | 11 | 22
  Not improved | 5 | 0
Statistical Analysis 1: Comparison: 'Hammock' Technique vs U-Method; The test applies to the number of participants improved; Test type: Superiority or Other; p = 0.0087, Fisher Exact

3. Secondary Outcome: Safety of the Sling.
Description: Safety of the sling was assessed with a record of perioperative and postoperative complications. The following are all the complications experienced with the TVT-SECUR for each technique, the 'Hammock' technique and the 'U-Method'.
Time Frame: 15 months
Population: The 'Hammock' technique, similar to the transobturator tape dissection, was used in the first 23 cases and the 'U-Method', similar to the retropubic tape dissection, in the last 25 cases. Interim analysis performed after 23 cases led us to change the technique to the 'U-Method'.
Measure: Number; unit: Participants
Groups:
- U-Method: The 'U-Method' is similar to the retropubic tape dissection.
Arm/Group | 'Hammock' Technique | U-Method
Number analyzed (Participants) | 25 | 23
Participants
  Perioperative urethral laceration | 0 | 1
  Postoperative vaginal erosions | 6 | 0
  Postoperative transient urinary retention | 0 | 2

ADVERSE EVENTS:
Arm/Group | TVT-SECUR

LIMITATIONS AND CAVEATS:
The single-surgeon single-center experience and the lack of objective outcome evaluation. A measurement bias of the 'U-Method' because of a learning curve for the cases using the 'Hammock' technique.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes